CLINICAL TRIAL: NCT01471808
Title: Effects of Oral Hypoglycemic Agents Combined With Short-term CSII on Glycemic Control in Newly-diagnosed Type 2 Diabetic Patients
Brief Title: Effects of Different Early Intensive Therapies on Long-term β-cell Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University Shenzhen Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Yanbing Li, the director of the endocrinology department of the First Affiliated Hospital of Sun Yat-sen University, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13560475186
Record Dates: First submitted 2011-11-08; First posted 2011-11-16 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- CSII (Active Comparator): continuous subcutaneous insulin infusion
  Interventions: Drug: CSII
- Metformin & Pioglitazone (Active Comparator): CSII combined with metformin and pioglitazone
  Interventions: Drug: CSII, Metformin, Pioglitazone
- Sitagliptin (Active Comparator): CSII combined with sitagliptin 100mg/d
  Interventions: Drug: CSII, Sitagliptin

INTERVENTIONS:
Drug: CSII — continuous subcutaneous insulin infusion for 2~4 weeks
  Arms: CSII
Drug: CSII, Metformin, Pioglitazone — CSII for 2~4 weeks combined with metformin 1.5g/d and pioglitazone 30mg/d for 3 months.
  Arms: Metformin & Pioglitazone
Drug: CSII, Sitagliptin — CSII for 2~4 weeks combined with sitagliptin 100mg/d for 3 months
  Arms: Sitagliptin

SUMMARY:
The purpose of this study is to investigate and evaluate the effects of different oral antihyperglycaemic agents combined with short-term continuous subcutaneous insulin infusion(CSII)(1.CSII alone; 2.metformin and pioglitazone combined with CSII; 3. sitagliptin combined with CSII) on long-term glycemic control and β-cell function in newly diagnosed type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes
* fasting blood glucose (FBG) level ranging from 7.0～16.7 mmol/L
* body mass index (BMI) ranging from21～35kg/m2
* Antihyperglycaemic and antihyperlipidemic medication-naive patients

Exclusion Criteria:

* having any severe acute or chronic diabetic complications
* renal dysfunction, blood creatinine≥150µmol/L
* blood aminotransferase level rising up(more than 2 times of the upper normal limit of ALT)
* • Any severe cardiac disease including congestive cardiac failure, unstable angina or myocardial infarct in 12 months
* chronic or acute pancreatic disease
* severe systematic diseases or malignant tumor
* female patients incline to be pregnant
* being treated with corticosteroid, immunosuppressing drugs or cytotoxic drugs
* poor compliance

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
proportions of 1 year remission of type 2 diabetes | 1 years
  the remission rate after short intensive therapy in newly diagnosed type 2 diabetic patients

SECONDARY OUTCOMES:
the effects of different interventions on β-cell function in newly-diagnosed type 2 diabetic patients | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Li, MD, Principal Investigator — Ministry of Education

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu L, Ke W, Wan X, Zhang P, Cao X, Deng W, Li Y. Insulin requirement profiles of short-term intensive insulin therapy in patients with newly diagnosed type 2 diabetes and its association with long-term glycemic remission. Diabetes Res Clin Pract. 2015 May;108(2):250-7. doi: 10.1016/j.diabres.2015.02.011. Epub 2015 Feb 21. PMID 25765670